CLINICAL TRIAL: NCT00553579
Title: The Relationship of Residence Time and Visual Effect of Optive and Systane in Dry Eye Subjects
Status: Completed | Type: Observational
Sponsor: Southern California College of Optometry at Marshall B. Ketchum University (Other)
Other Study IDs: SCCO2-2241
Record Dates: First submitted 2007-11-01; First posted 2007-11-05 (Estimated); Last update posted 2008-05-20 (Estimated); Status verified 2008-05

CONDITIONS: Dry Eye Disease
Keywords: contrast sensitivity, retention time
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- DE: All subjects will have clinically significant dry eye.

SUMMARY:
The benefits of artificial tears to relieve dry eye symptoms include, but are not limited to: stabilizing the tear film layer, fluid supplement action, improving visual acuity, and comfort. Studies have found a relationship between some of these benefits. For example, stabilization of the tear film is important not only to increase the tear break up time (TBUT), but is key in improving and maintaining visual acuity. These studies have alluded to the fact that there may or may not be a relationship between residence time and visual performance. Viscosity is one reason behind the uncertainty. Some solutions contain polymers which influence the ocular surface when contacted. This can impact residence time and ultimately visual performance. No prior research has explored the direct relationship between residence time and visual performance.

Residence time refers to the duration at which the artificial tear resides on the eye. Methods have been developed to assess residence time by admixing fluorescent tracers to the solution and then measuring the amount of fluorescence over time. The caveat to methods using certain tracers has lead to uncertainty in elimination measurements due to corneal penetration or differing molecular weights (MW) from the active vehicle ingredient in the solution. For example, low-MW tracers can be eliminated at a different rate than higher-MW polymers. In addition, the low-MW tracers may be able to penetrate the corneal epithelium giving a false pre-corneal residence time. Meadows, Paugh, Joshi, and Mordaunt addressed this issue by developing a technique using a polymer which did not penetrate the cornea and had the same MW as the active ingredient in the solution FITC-dextran. Based on the assumption that similar weights are eliminated at the same rate, this technique has shown to be more economic, manageable, and amendable than previous procedures measuring residence time.

Any ophthalmic drop has the potential to impact visual acuity upon instillation due to the effect it has on the tear layer components. Studies have observed that taking artificial tears continuously over time tends to stabilize the tear layer thus minimizing the immediate drop in contrast sensitivity upon instillation. Measuring the visual effect of artificial tears, using contrast sensitivity as a measure, provides valuable information about the therapeutic effect of artificial tears that are meant to stabilize the tear film, thus improving visual acuity in dry eye patients.

But what about the patient? There is a difference between residence time and retention of effect- which is often what matters the most for patients. Retention of effect refers to the beneficial effect of the drop. Currently there is no real measure of retention of effect. Doctors can assess the tear film objectively, but there have been no strong correlations between subjective dry symptoms and tear film stability. A possible reason for the lack of correlation may be due to the fact that subjectivity is difficult to quantify. However, scales like the Visual Analog Scale (VAS) and Numerical Rating Scale (NRS) have been established in an attempt to quantify subjective experiences such as visual quality. We will be using the NRS to gauge the comfort of the drop upon the initial application to get a general idea of the comfort the drop provides to the user.

Although there have been several studies done on residence time and visual effect of ophthalmic formulations separately, there is no current research correlating these two aspects of therapeutic efficacy. This study will be the first to concurrently investigate residence time (using FITC-dextran) and visual effect of an ophthalmic formulation.

ELIGIBILITY:
Inclusion Criteria:

* There are no requirements as to subject race, gender or occupation. All subjects must meet the following criteria:

  * The informed consent document must be read, signed and dated by the subject or legally authorized representative before conducting any procedures. Additionally, the informed consent document must be signed and dated by the individual obtaining consent of the subject.
  * Adult subjects, > age 18 years, with mild-to-moderate dry eye. Criteria for the diagnosis must include two of the three following characteristics as demonstrated at the Eligibility Visit:
  * Composite symptom score of ≥ 7 on the Schein Questionnaire:
  * Sodium Fluorescein (NaFl) Tear Break-Up Time ≤ 7 seconds in either (worse) eye
  * Cumulative Sodium Fluorescein (NaFl) Corneal Staining ≥ 4 in either (worse) eye on a 0-20 point scale (corresponds to ≥ 3 on a 0-15 scale).
  * Able and willing to follow study instructions.
  * Subjects must have best corrected visual acuity of 20/25 or better in each eye as assessed using an ETDRS chart.

Exclusion Criteria:

* Subjects demonstrating any medical condition that may affect the results of this study will NOT be enrolled. The following are specific conditions that exclude subjects from enrollment in this study.

  * History or evidence of ocular or intraocular surgery in either eye within the past six months. LASIK and other keratorefractive procedure patients can qualify if the most recent surgery or enhancement was 12 or more months prior.
  * History or evidence of serious ocular trauma in either eye within the past six months.
  * History of hypersensitivity to any component of the study medications: History of hypersensitivity to any component of Optive® Artificial Tears, Systane® Artificial Tears, diagnostic dyes sodium fluorescein and fluorescein isothiocyanate dextran.
  * History or evidence of epithelial herpes simplex keratitis (dendritic keratitis); vaccinia, active or recent varicella, viral disease of the cornea and/or conjunctiva; chronic bacterial disease of the cornea and/or conjunctiva; mycobacterial infection of the eye; and/or fungal disease of the eye.
  * Use of concomitant topical ocular medications during the study period.
  * Subjects using systemic steroids, immunosuppressive agents and/or anti-cholinergics (e.g. cold and allergy medications, tricyclic antidepressants) for treatment of autoimmune connective tissue disease may not be enrolled in the study if they have not been on a stable dosing regimen for a minimum of 30 days prior to the Eligibility Visit. In addition, the dosing regimen must remain stable throughout the study period.
  * Ocular conditions such as conjunctival infections, or iritis.
  * Individuals unwilling to discontinue contact lens wear for 2 days prior to each visit during the study period.
  * Participation in an investigational drug or device study within 30 days of entering this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The subjects for this investigation will be sourced from an existing, secure dry eye subject database. These subjects will have been screened for dry eye using a consistent protocol (Diagnostic monograph, J. Paugh, January 2007). Subjects who have taken part in a prior study undergoing this same eligibility visit protocol within the past 18 months will not be required to repeat the visit.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Estimated)
Dates: Start 2007-06; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
The principal outcome parameters will be gross residence time in minutes and the effect on contrast sensitivity time in minutes. | 1 hour

SECONDARY OUTCOMES:
A secondary outcome variable will be the comfort value (NRS) of the initial drop application. | 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: William Ridder, OD, PhD, Principal Investigator — Southern California College of Optometry at Marshall B. Ketchum University
Locations (1):
- Southern California College of Optometry, Fullerton, California, United States